CLINICAL TRIAL: NCT05664737
Title: A Phase 2, Study for the Treatment of Anemia With Alpha (α)-Thalassemia to Determine the Efficacy and Safety of Luspatercept (BMS-986346/ACE-536) in Adults and Evaluate the Safety and Pharmacokinetics in Adolescents
Brief Title: A Study to Determine the Efficacy and Safety of Luspatercept in Adult Participants and to Evaluate the Safety and Pharmacokinetics in and Adolescent Participants With Alpha (α)-Thalassemia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CA056-015; 2022-502328-35 (Other: EU CTR)
Record Dates: First submitted 2022-12-09; First posted 2022-12-27 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Anemia
Keywords: Luspatercept; BMS-986346; ACE-536; α-thalassemia; Alpha Thalassemia; Reblozyl; Transfusions; Non-transfusion dependent; RBC transfusion dependent
MeSH Terms: conditions — Anemia; alpha-Thalassemia | interventions — luspatercept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Transfusion Dependent (TD): Luspatercept + Best supportive care (BSC) (Experimental)
  Interventions: Biological: Luspatercept
- Adult TD Cohort: Placebo + BSC (Placebo Comparator)
  Interventions: Drug: Placebo
- Non-transfusion Dependent (NTD): Luspatercept + BSC (Experimental)
  Interventions: Biological: Luspatercept
- Adult NTD Cohort: Placebo + BSC (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: Luspatercept — Specified dose on specified days
  Other Names: BMS-986346; ACE-536; REBLOZYL
  Arms: Non-transfusion Dependent (NTD): Luspatercept + BSC; Transfusion Dependent (TD): Luspatercept + Best supportive care (BSC)
Drug: Placebo — Specified dose on specified days
  Arms: Adult NTD Cohort: Placebo + BSC; Adult TD Cohort: Placebo + BSC

SUMMARY:
The purpose of the study is to evaluate the efficacy and safety of luspatercept plus best supportive care (BSC) vs placebo plus BSC on anemia in adult participants with α-thalassemia hemoglobin H (HbH) disease and determine the safety and drug levels in adolescent participants.

ELIGIBILITY:
Key Inclusion Criteria:

* Adult participant≥ 18 years with documented diagnosis of A-Thal HbH disease with Transfusion dependence defined as:.

  1. TD participant: ≥ 6 RBC units during the 24 weeks prior to randomization.
  2. NTD participant:< 6 RBC units during the 24 weeks prior to randomization(transfusion due to conditions other than A-Thal will not be considered)and, RBC transfusion-free during at least 8 weeks prior to randomization(unless transfusion was required to treat an acute medical condition other than A-Thal) and, mean baseline Hb ≤ 10 g/dL, based on a minimum of 2 measurements ≥ 1 week apart within 4 weeks prior to randomization; hemoglobin values within 21 days post-transfusion will be excluded.
* Adult participant has Eastern Cooperative Oncology Group (ECOG) 34 score of 0 or 1.
* Adolescent participant 12 years to < 18 years with documented diagnosis of A-Thal HbH disease with transfusion dependence defined as:.

  1. TD participant: ≥ 4 RBC events during the 24 weeks prior to enrollment and, no transfusion-free period for > 56 days during the 24 weeks prior to enrollment. Participants must have a history of regular transfusions for at least 2 years.
  2. NTD participant:< 4 RBC events during the 24 weeks prior to enrollment and RBC transfusion-free during at least 8 weeks prior to enrollment and, mean baseline Hb ≤ 10 g/dL, based on a minimum of 2 measurements ≥ 1 week apart within 4 weeks prior to enrollment, hemoglobin values within 21 days post-transfusion will be excluded.
  3. Participant has Karnofsky (age ≥16 years) or Lansky (age < 16 years) performance status score ≥ 50 at screening.

Key Exclusion Criteria:

* Medical Conditions: Diagnosis of A-ThalTrait, Hb Bart hydrops, ATRx A-Thal, hemoglobin S/β-thalassemia, myelodysplasia subtype anemia, or with HbE homozygous beta gene mutation. Anemia related to nutritional deficiency, anemia of chronic disease, autoimmune hemolytic anemia, or any other hemolytic anemias. Undergone episodes of hemolysis not related to A-Thal within the 8 weeks prior to randomization.
* Participant has deep vein thrombosis (DVT), stroke or other thromboembolic event(s) (except clogged indwelling catheter) requiring medical intervention ≤ 24weeks prior to randomization.
* Participant has uncontrolled hypertension. Controlled hypertension for this protocol is considered: blood pressure value corresponding to ≤Grade 1 according to NCI CTCAE Version 5.0. with or without pharmacological treatment.
* Reproductive Status: Women who are pregnant, plan to get pregnant during the study, or who are breastfeeding.
* Prior/Concomitant: Undergone HSCTs or gene therapy (candidates for HSCT or gene therapy with waiting period of ≥ 12 months are eligible).
* Use of hydroxyurea treatment ≤ 12 weeks prior to enrollment for NTD participants and ≤ 24 weeks for TD participants.
* Participant who has extramedullary hematopoiesis (EMH) complications requiring treatment to control the growth of EMH mass(es) during the screening period.
* Any medical or psychiatric condition (including active infections, recent surgery, sequelae of diseases or interventions, clinically significant laboratory abnormalities or concurrent treatment) that in the opinion of the investigator would put the participant at unacceptable risk of participating in the study or that could affect interpretability of data.
* Other protocol-defined inclusion/exclusion criteria apply.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 249 (Estimated)
Dates: Start 2022-12-09 (Actual); Primary Completion 2027-07-16 (Estimated); Study Completion 2034-08-14 (Estimated)

PRIMARY OUTCOMES:
Number of participants with ≥ 50% reduction from baseline in RBC transfusion burden with a reduction of at least 2 units during any continuous 12 weeks during Week 13-48 compared to 12-week interval immediately prior to date of first dose | Up to Week 48
  Adult TD Cohort
Number of participants with an increase from baseline of ≥ 1.0 grams (g)/decilitre (dL) in mean hemoglobin (Hb) values over the continuous 12-week interval from Week 13 to Week 24 in the absence of RBC transfusion | Up to Week 24
  Adult NTD Cohort
Dose-limiting toxicities (DLTs) defined as observance of ≥ Grade 3-related hemolytic crises or ≥ Grade 3-related event outside of the known safety profile occurring within the 21 days from their first dose of study therapy | Up to Week 3
  Adolescent TD and NTD Cohorts
Number of participants with adverse events (AEs) | Up to 8.5 years
  Adolescent TD and NTD Cohorts
Pharmacokinetics (PK): Serum concentration of Luspatercept | Up to Week 102
  Adolescent TD and NTD Cohorts

SECONDARY OUTCOMES:
Number of participants with ≥ 33% reduction from baseline in RBC transfusion burden with a reduction of at least 2 units during any continuous 24-week interval on treatment compared to 24-week interval immediately prior to date of first dose | Up to Week 108
  Adult TD Cohort
The longest duration with ≥ 50% reduction from baseline in RBC transfusion burden with a reduction of at least 2 units | Up to Week 108
  Adult TD Cohort
Number of RBC transfusion units from week 1 to week 48 | Up to Week 48
  Adult and Adolescent TD Cohorts
Change from baseline in hemoglobin in the absence of transfusion at Week 24 | Up to Week 24
  Adult and Adolescent NTD Cohorts
The longest duration of an increase from baseline of ≥ 1.0 g/dL in mean hemoglobin values starting from Week 13 in the absence of transfusion | Up to Week 108
  Adult NTD Cohort
Time Duration with an increase from baseline of ≥ 1.0 g/dL in hemoglobin values in the absence of transfusion within 48 weeks | Up to Week 48
  Adult NTD Cohort
Number of participants with an increase from baseline of ≥1.0 g/dL in mean Hb values over the continuous 12- week interval in the absence of transfusion | Up to Week 24
  Adult NTD Cohort
≥ 3 Increase from Baseline in Functional Assessment of Cancer Therapy Anemia Fatigue Subscale (FACT-An FS) Score from Baseline to the period from Week 13 to Week 24 | Up to Week 24
  Adult NTD Cohort
Number of participants with AEs | Up to 5 years
  Adult and Adolescent TD and NTD Cohorts
Number of participants with laboratory abnormalities | Up to 5 Years
  Adult TD and NTD Cohorts
Number of participants with immunogenicity | Up to 5 Years
  Adult TD and NTD Cohorts
Number of participants with ≥ 50% reduction from baseline in RBC transfusion burden during any continuous 24-week interval within 48 weeks compared to the 24-week interval immediately prior to the date of first dose | Up to Week 48
  Adult TD Cohort
Number of participants with ≥ 33% reduction from baseline in RBC transfusion burden during any continuous 12-week interval compared to the 12-week interval immediately prior to the date of first dose | Up to Week 108
  Adult TD Cohort
Number of participants with ≥ 33% reduction from baseline in RBC transfusion burden from Week 13 to Week 24 and Week 37 to Week 48 compared to the 12-week interval immediately prior to the date of first dose | Up to Week 48
  Adult TD Cohort
Number of participants with ≥ 33% reduction from baseline in RBC transfusion burden from Week 1 to Week 24 and Week 25 to Week 48 compared to the 24-week interval immediately prior to the date of first dose | Up to Week 48
  Adult TD Cohort
Number of participants with ≥ 50% reduction from baseline in RBC transfusion burden from Week 13 to Week 24 and Week 37 to Week 48 compared to the 12-week interval immediately prior to the date of first dose | Up to Week 48
  Adult TD Cohort
Number of participants with ≥ 50% reduction from baseline in RBC transfusion burden from Week 1 to Week 24 and Week 25 to Week 48 compared to the 24-week interval immediately prior to the date of first dose | Up to Week 48
  Adult TD Cohort
Change from baseline in total RBC units transfused from Week 1 to Week 24, Week 25 to Week 48, and Week 1 to Week 48 | Up to Week 48
  Adult TD Cohort
The longest duration of RBC transfusion-free period for participants who achieve transfusion-free period of ≥ 12 weeks | Up to Week 108
  Adult TD Cohort
The longest duration of reduction in transfusion burden for participants who achieve a response (rolling 12-week and 24-week response, both for ≥ 33% and ≥ 50% reduction) | Up to Week 108
  Adult TD Cohort
Time from first dose to first day of response (rolling 12-week and 24-week response, both for ≥ 33% and ≥ 50% reduction) | Up to Week 108
  Adult TD Cohort
Change from baseline in number of transfusion events at Week 48 | Up to Week 48
  Adult TD Cohort
Number of participants who achieve RBC transfusion-free period of any continuous ≥ 12 weeks during treatment | Up to Week 108
  Adult and Adolescent TD and NTD Cohorts
Number of participants who achieve RBC transfusion-free period of any continuous ≥ 24 weeks during treatment | Up to Week 108
  Adult and Adolescent TD and NTD Cohorts
Time to first transfusion | Up to Week 108
  Adult and Adolescent NTD Cohorts
Number of transfusions | Within 48 Weeks
  Adult NTD Cohort
Number of transfusion visits/units | Within 48 Weeks
  Adult NTD Cohort
Change from baseline in mean hemoglobin values over the continuous 12-week interval from Week 13 to Week 24 and Week 37 to Week 48 in the absence of transfusions | Up to Week 48
  Adult TD and NTD Cohorts
Number of participants achieving an increase from baseline of ≥1.0g/dL or ≥1.5g/dL in mean Hb values in absence of transfusions from Week 13 to Week 24, Week 37 to Week 48 and during any continuous 12-week window within 24 weeks and 48 weeks | Up to Week 48
  Adult NTD Cohort
Time from first to last Hb measurement with increase from baseline by ≥ 1.0 g/dL | Up to Week 108
  Adult NTD Cohorts
Time to the first increase from baseline of ≥ 1.0 g/dL in mean Hb value | Up to Week 48
  Adolescent NTD Cohort
Number of participants who achieve an increase in mean Hb of >10g/dL values during any continuous 12-week and 24-week interval within 48 weeks in the absence of transfusions | Up to Week 48
  Adult NTD Cohort
Change from baseline in self-reported health-related quality of life (HRQoL) assessed by physical component summary (PCS) and mental component summary (MCS) of 36-item short-form health survey version2 (SF-36v2) at Week 24 and Week 48 | Up to Week 48
  Adult TD and NTD Cohorts
Change from baseline in non-transfusion dependent β-thalassemia patient-reported outcome (NTDT-PRO) Tiredness/weakness (T/W) and shortness of breath (SoB) domain scores from Week 13 to Week 24 and from Week 37 to Week 48 | Up to Week 48
  Adult NTD Cohort
Change from baseline in FACT-An FS Score at Week 24 and Week 48 | Up to Week 48
  Adult NTD Cohort
Change from baseline in Functional Assessment of Cancer Therapy Anemia Anemia Subscale (FACT-An AS) at Week 24 and Week 48 | Up to Week 48
  Adult NTD Cohort
Number of participants with at least one hemolytic crisis | Up to Week 108
  Adult TD and NTD Cohorts
Rate of hemolytic crises | Up to Week 108
  Adult TD and NTD Cohorts
Time to first hemolytic crisis | Up to Week 108
  Adult TD and NTD Cohorts
Time to second hemolytic crisis | Up to Week 108
  Adult TD and NTD Cohorts
Change from baseline in hemolysis markers at Week 24 and Week 48 | Up to Week 48
  Adult TD and NTD Cohorts:
Change from baseline in the 6-minute walk test (6MWT) distance at Week 24 and Week 48 | Up to Week 48
  Adult NTD Cohort
Pharmacokinetics (PK): Serum concentration of Luspatercept | Up to Week 108
  Adult and Adolescent TD and NTD Cohorts
Percent Change from Baseline in Biomarkers for Erythropoiesis at Week 84 | Baseline, Week 84
  Adult TD and NTD Cohorts
  The biomarkers for erythropoiesis to be evaluated include Hb variants including hemoglobin H (HbH), sTfR1, erythropoietin (EPO), growth differentiation factor (GDF11), GDF8, GDF15. The change will be measured as a percentage of change from baseline for all the biomarkers.
Percent Change from Baseline in Biomarkers and Parameters for Iron Homeostasis at Week 84 | Baseline, Week 84
  Adult TD and NTD Cohorts
  The biomarkers and parameters for iron homeostasis to be evaluated include hepcidin, erythroferrone (ERFE), serum ferritin, liver iron concentration (LIC), myocardial iron, iron chelation therapy (ICT).
  The change will be measured as a percentage of change from baseline for all the biomarkers.
Change in mean corpuscular volume (MCV) at Week 48 | Baseline, Week 48
  Adult TD and NTD Cohorts
Change in mean corpuscular hemoglobin (MCH) at Week 48 | Baseline, Week 48
  Adult TD and NTD Cohorts
Change in nucleated red blood cells (nRBC) at Week 48 | Baseline, Week 48
  Adult TD and NTD Cohorts
Change in red blood cells (RBC) at Week 48 | Baseline, Week 48
  Adult TD and NTD Cohorts
The longest duration with reduction from baseline in the RBC transfusion burden | Up to Week 48
  Adolescent TD Cohort
The number of participants with ≥ 50% reduction from baseline in RBC transfusion burden during an continuous 12 weeks during Weeks 13-48 | Up to Week 48
  Adolescent TD Cohort
The number of participants with ≥ 33% reduction from baseline in RBC transfusion burden during an continuous 24 weeks | Up to Week 48
  Adolescent TD Cohort
Number of participants achieving an increase from baseline of ≥1.0g/dL in mean Hb values in absence of transfusions from Week 13 to Week 24 | Up to Week 24
  Adolescent NTD Cohort
Cumulative time (in weeks) with an increase from baseline of ≥1.0g/dL in mean Hb values in absence of RBC transfusions within 48 weeks | Up to Week 48
  Adolescent NTD Cohort
Number of participants who achieve an increase in mean Hb of >10g/dL values during any continuous 12-week interval during week 13 to week 48 in the absence of transfusions | Up to Week 48
  Adolescent NTD Cohort
The longest duration with an increase from baseline of ≥1.0g/dL in mean Hb values in absence of transfusions | Up to Week 48
  Adolescent NTD Cohort
Number of participants with antidrug antibody (ADA) | Up to Week 48
  Adolescent TD and NTD Cohorts
Mean change in biomarkers for hemolysis | Up to Week 48
  Adolescent TD and NTD Cohorts
  Biomarkers for hemolysis to be evaluated include total/direct/indirect bilirubin, serum lactate dehydrogenase (sLDH), haptoglobin, reticulocytes and nucleated red blood cells, reticulocyte production index (RPI), and urinary urobilinogen
Mean change in biomarkers and parameters for iron homeostasis | Up to 1 Year
  Adolescent TD and NTD Cohorts
  The biomarkers and parameters for iron homeostasis to be evaluated include serum ferritin, LIC, myocardial iron concentration (MIC), ICT, myocardial T2(TD participants), and extramedullary hematopoiesis (EMH) mass(es) when present (NTD participants)
Hematologic assessments | Up to Week 48
  Adolescent TD and NTD Cohorts
  The hematologic assessments to be evaluated are red blood cell count, hemoglobin, hematocrit, reticulocyte count, nucleated red blood cell count, platelet count, mean cell volume, mean cell hemoglobin, mean corpuscular hemoglobin concentration, red blood cell distribution width, red blood cell morphology, and globin precipitates
The change from baseline in the number of health care resource utilization (HCRU) | Up to Week 48
  Adolescent TD and NTD Cohorts
Mean change from baseline in Pediatric Quality of Life Inventory (PedsQL) domain scores | Up to Week 48
  Adolescent TD and NTD Cohorts
Mean change from baseline EQ-5D-5L utility index | Up to Week 48
  Adolescent TD and NTD Cohorts
Mean change from baseline visual analogue scale (VAS) scores | Up to Week 48
  Adolescent TD and NTD Cohorts

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (36):
- Local Institution - 0008, Halifax, Nova Scotia, Canada
- China (11):
  - Sun Yat-sen Memorial Hospital, Sun Yat-Sen University, Guangzhou, GD
  - Nanfang Hospital of Southern Medical University, Guangzhou, GD
  - The First People's Hospital of Foshan, Foshan, Guangdong
  - Maoming People's Hospital, Maoming Shi, Guangdong
  - Shenzhen Second People's Hospital, Shenzhen Shi, Guangdong
  - Liuzhou People's Hospital, Liuchow, Guangxi
  - People's Liberation Army The 923rd Hospital, Nanning, GX
  - Local Institution - 0011, Haikou, Hainan
  - Local Institution - 0012, Kunming, Yunnan
  - Hainan General Hospital, Haikou
  - The First Affiliated Hospital of Guangxi Medical University, Nanning
- Greece (5):
  - Local Institution - 0005, Thessaloniki, B
  - Local Institution - 0007, Larissa, E
  - Local Institution - 0018, Rio, G
  - Local Institution - 0006, Athens
  - Local Institution - 0009, Goudi
- Hong Kong (2):
  - Local Institution - 0025, Hong Kong, HK
  - Local Institution - 0024, Hong Kong Island
- Italy (5):
  - Local Institution - 0022, Cagliari, CA
  - Local Institution - 0026, Genova, GE
  - Local Institution - 0020, Orbassano, TO
  - Local Institution - 0028, Napoli
  - "Universita degli Studi della Campania ""Luigi Vanvitelli"" - AOU - Clinica Pediatrica", Napoli
- Malaysia (2):
  - Hospital Tunku Azizah, Kuala Lumpur, WP
  - Hospital Sultanah Aminah, Johor Bahru
- Saudi Arabia (2):
  - Local Institution - 0035, Al-Ahsa
  - King Saud University (KSU) - College of Medicine, Riyadh
- KK Women's and Children's Hospital, Singapore, Singapore
- Taiwan (3):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City, KHH
  - National Taiwan University Hospital, Nan Gang Qu, TPE
  - China Medical University Hospital, Taichung, TXG
- Thailand (2):
  - Siriraj Hospital, Bangkok Noi, Bangkok
  - Naresuan University Hospital, Mueang Phitsanulok
- Turkey (Türkiye) (2):
  - Hacettepe Üniversitesi Tıp Fakültesi, Altındağ
  - Istanbul Universitesi - Istanbul Tip Fakultesi (ITF) Hastanesi, Topkapı

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myer Squibb's data sharing policy and process can be found at https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html

REFERENCES:
- [Derived] Diamantidis MD, Pitsava S, Zayed O, Argyrakouli I, Karapiperis K, Chatzoulis C, Alexiou E, Manafas A, Tsangalas E, Karakoussis K. Concomitant Presence of Hb Agrinio and - -Med Deletion in a Greek Male Patient with Hemoglobinopathy H: More Severe Phenotype and Literature Review. Hematol Rep. 2023 Aug 8;15(3):483-490. doi: 10.3390/hematolrep15030050. PMID 37606495
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT05664737.html